CLINICAL TRIAL: NCT00612716
Title: Unrelated or Partially Matched Allogeneic Donor Stem Cells for Lymphoma, Myeloma, and Chronic Lymphocytic Leukemia
Brief Title: Donor Stem Cell Transplant in Treating Patients With Previously Treated Lymphoma, Multiple Myeloma, or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1999LS060; 9909M18181 (Other: IRB, University of Minnesota); UMN-MT1999-14 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2008-02-09; First posted 2008-02-12 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; recurrent adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage II adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage II adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; stage I adult lymphoblastic lymphoma; stage II adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent childhood anaplastic large cell lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; Burkitt lymphoma; recurrent childhood small noncleaved cell lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Hodgkin Disease; Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating | interventions — Busulfan; Cyclophosphamide; Cord Blood Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Transplantation, Homologous; Bone Marrow Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Transplantation (Experimental): Patients receiving total body irradiation, stem cell infusion (allogeneic)transplantation using unrelated or partially matched allogeneic marrow or cord blood donors, busulfan, and cyclophosphamide.
  Interventions: Drug: busulfan; Drug: cyclophosphamide; Biological: Stem cell infusion; Radiation: Total body irradiation

INTERVENTIONS:
Drug: busulfan — For those not eligible for total body irradiation: busulfan 4 mg/kg/day orally (1 mg/kg orally every 6 hrs) on Days -9 through -6.
  Other Names: Busulfex
Drug: cyclophosphamide — Cyclophosphamide 60 mg/kg/day on days -7 and -6. For patients not eligible for total body irradiation: cytoxan 50 mg/kg intravenously (IV) on days -5 through -2.
  Other Names: Cytoxan
Biological: Stem cell infusion — Infused on Day 0
  Other Names: umbilical cord blood transplantation; hematopoietic stem cell transplantation; allogeneic transplantation; bone marrow transplantation
Radiation: Total body irradiation — 165 cGy morning and evening on days -4 through -1.
  Other Names: TBI

SUMMARY:
RATIONALE: Giving chemotherapy, such as cyclophosphamide and busulfan, and total-body irradiation before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells from bone marrow or umbilical cord blood may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving methotrexate and cyclosporine after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well a donor stem cell transplant works in treating patients with previously treated lymphoma, multiple myeloma, or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if allogeneic stem cell transplantation using unrelated matched or related haploidentical donor bone marrow or unrelated matched cord blood results in timely, complete, and durable engraftment in patients with previously treated lymphoma, multiple myeloma, or chronic lymphocytic leukemia.
* Determine the incidence and grade of acute and chronic graft-versus-host disease in patients treated with this regimen.
* Determine if the augmented graft-versus-tumor effect accompanying unrelated or partially matched donor allogeneic transplant reduces the incidence of relapse in these patients.

OUTLINE:

* Preparative regimen: Patients receive cyclophosphamide IV over 2 hours on days -7 and -6 and undergo total-body irradiation (TBI) twice daily on days -4 to -1. Patients who are unable to undergo TBI receive busulfan IV or orally 4 times daily on days -9 to -6 and cyclophosphamide IV over 2 hours on days -5 to -2.
* Stem cell transplantation: All patients undergo unrelated matched bone marrow or umbilical cord blood transplantation or partially matched related allogeneic bone marrow transplantation on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive GVHD prophylaxis comprising methotrexate and cyclosporine. Patients may be enrolled in other protocols directed towards GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Donors will be <55 years of age and in good health as approved by the National Marrow Donor Program (NMDP) donor and collection centers. Related donors will be < 70 years of age.
* Recipients will be <55 years, will have satisfactory organ function (excluding bone marrow) and will have a Karnofsky activity assessment >90% and will have:

  * Creatinine <2.0 mg/dl.
  * Bilirubin, Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2 x normal.
  * Pulmonary function test and Carbon Monoxide Diffusing Capacity (DLCO) > 50% of normal.
  * Multi Gated Acquisition Scan (MUGA) >45% injection fraction.
* Recipients with unrelated donor matched at the HLA A, B, DRBI loci, or if < 35 years mismatched at a single HLA A or B, or DRBI locus.
* Umbilical cord blood (5) used as an unrelated stem cell source will provide > 2.0 x 10^7 cells/kg and will be matched at 4 - 6 of 6 HLA A, B, and DRBI loci. Cord blood grafts may include a single or pair of cord units depending on the cell dose.
* Partially matched related donors will be at least haploidentical (matched at >3 of 6 HLA A, B, DRB1 loci).
* Recipients will fall under one of the following disease categories

  * Chronic lymphocytic leukemia -- must have all three:

    * Rai Stage III/IV
    * Progression after previous Complete Response (CR) or Partial Response (PR) including purine antagonist (i.e. fludarabine).
    * Recent chemotherapy responsiveness
  * Advanced non-Hodgkin's lymphoma(NHL).

    * Low-grade NHL (Working Formulation A, B, C) following progression after initial therapy if asymptomatic at diagnosis (>CR2, >PR2; response duration < 1 year from last therapy) or if no CR was achieved (>PR1). At least one prior therapy of intermediate intensity (e.g. CHOP).
    * Mantle zone lymphoma after any progression following initial therapy (>CR1, > PR1). At least one prior therapy of intermediate intensity (e.g. CHOP).
    * Intermediate grade lymphoma (>PR2). Response duration <1 year from prior therapy.
    * High-grade Non-Hodgkin's Lymphoma (NHL) (IWF H, I, J) after initial therapy if >stage III at diagnosis; after any progression even if localized (stage I, II) at diagnosis with prior response duration < 1 year.
    * Recent chemotherapy responsiveness after treatment with > 3 intermediate intensity regimens.
  * Advanced Hodgkin's disease beyond PR2 (>CR3, >PR3).

    * Recent chemotherapy responsiveness
  * Multiple Myeloma (>CR2, >PR2) or after initial therapy if no prior PR.

    * Recent chemotherapy responsiveness
* Recipients will sign informed consent approved by the Committee on the Use of Human Subjects at the University of Minnesota.

Exclusion Criteria:

* No available histocompatible related donor; 2nd bone marrow transplant (BMT), HIV-1 positive; active uncontrolled infection; or resistant malignancy.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 1999-10-06 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Weisdorf, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allogeneic Transplantation
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Engraftment Failure
Description: Graft failure is defined as not accepting donated cells. The donated cells do not make the new white blood cells, red blood cells and platelets.
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Number of Participants With Neutrophil Engraftment
Description: Time to 1st 3 consecutive days with absolute neutrophil count (ANC) > 5 x 10^8/L and percentage of patients with neutrophil recovery by day 42 (Cumulative incidence).
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 6
Participants | 5

3. Primary Outcome: Number of Participants With Platelet Engraftment
Description: Time to platelets > 20,000 (first of 3 consecutive days) with no platelet transfusions for seven days and percentage of patients with platelet engraftment >50,000 by day 100.
Time Frame: Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 6
Participants | 2

4. Primary Outcome: Number of Participants With Grade 3-4 Acute Graft-versus-host Disease
Description: Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 6
Participants | 3

5. Primary Outcome: Number of Participants With Persistence Disease
Description: the return of disease after its apparent recovery/cessation.
Time Frame: 3 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 6
Participants | 1

6. Primary Outcome: Number of Participants With Relapse of Malignancy
Description: the return of disease after its apparent recovery/cessation.
Time Frame: 3 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 6
Participants | 1

7. Primary Outcome: Number of Participants With 1 Year Overall Survival
Description: The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease, such as cancer. Also called survival rate.
  Overall survival will be defined as time from date enrollment to date of death or censored at the date of last documented contact for patients still alive.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 6
Participants | 2

8. Primary Outcome: Number of Participants With 2 Year Overall Survival
Description: as for outcome 7
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 6
Participants | 1

9. Secondary Outcome: Number of Participants With of Chronic GVHD.
Description: Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Allogeneic Transplantation
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Transplantation (N=6)
Primary graft failure (Injury, poisoning and procedural complications) | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) — primary cause graft failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Transplantation (N=6)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Platelet refractory (Blood and lymphatic system disorders) | 1 (1)
Abnormal bilirubin (Infections and infestations) | 3 (6)
Active Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6)
Acute respiratory distress syndorme (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute sinusitis (Reproductive system and breast disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorder, other (Cardiac disorders) | 1 (1)
Cyclosporine renal dysfunction (Renal and urinary disorders) | 2 (2)
Dialysis (Renal and urinary disorders) | 3 (3)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1)
Drug toxicity (Skin and subcutaneous tissue disorders) | 2 (2)
Duodenal capillary congestion (Blood and lymphatic system disorders) | 1 (1)
Elevated Partial Thromboplastin Time (Investigations) | 1 (1)
Embolization of uterine artery (Renal and urinary disorders) | 1 (1)
Epileptic episode (Nervous system disorders) | 1 (1)
GI bleeding (Gastrointestinal disorders) | 4 (5)
Graft vs host disease (Immune system disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 4 (5)
Hemolytic uremia (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Hypogonadism (Reproductive system and breast disorders) | 2 (2)
Hypokalemic (Investigations) | 1 (1)
Hypomagnesmia (Investigations) | 1 (1)
Increased creatinine (Renal and urinary disorders) | 2 (2)
Infection (Infections and infestations) | 5 (80)
Intubation (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Learning Dysfunction (Nervous system disorders) | 1 (1)
muscle disorder other (Musculoskeletal and connective tissue disorders) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Neurotoxicity (Nervous system disorders) | 2 (2)
Pancytopenic (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (5)
Renal failure (Renal and urinary disorders) | 4 (4)
Seizure (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septicemia (Infections and infestations) | 1 (1)
Subarachoid bleed (Blood and lymphatic system disorders) | 1 (1)
Thrombosis (Blood and lymphatic system disorders) | 1 (2)
Uremic platelet dysfunction (Blood and lymphatic system disorders) | 1 (2)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1)
Vascular disorder, other (Blood and lymphatic system disorders) | 1 (1)
Veno occulisive disease (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-05-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT00612716/Prot_SAP_000.pdf